CLINICAL TRIAL: NCT03898843
Title: Assisted Animal Therapy in a French Intensive Care Unit (ICU): An Open Randomized Study
Brief Title: Assisted Animal Therapy: ReAnimal
Acronym: ReAnimal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrollment and logistical problems
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0804; 2018-A02789-46 (Other: ID-RCB)
Record Dates: First submitted 2019-03-27; First posted 2019-04-02 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Mood Disorders; Post Traumatic Stress Disorder
Keywords: Animal assisted therapy; Intensive Care Unit; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Stress Disorders, Post-Traumatic | interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal assisted therapy group (Experimental): Patients included in this arm will have animal assisted therapy session in a specific room outside of the ICU. They will also have blood sampling for multidrug resistant bacteria screening and will answer to questionnaires
  Interventions: Other: Animal assisted therapy; Biological: Nasal swab sampling; Behavioral: STAI-Y and POMS Questionnaires; Procedure: physiological parameters measure; Other: Visual Analog Scale (VAS); Behavioral: Impact of Event Scale - Revised (IES-R); Behavioral: satisfaction questionnaire; Biological: Rectal swab sampling
- Control Group (Active Comparator): Patients included in this arm will have a "sham session" : they will leave their hospital bedroom, to go in the AAT session room. There, no specific activity is planned. After 20 minutes, the patient will go back to his room. They will also have blood sampling for multidrug resistant bacteria screening and will answer to questionnaires
  Interventions: Biological: Nasal swab sampling; Behavioral: STAI-Y and POMS Questionnaires; Procedure: physiological parameters measure; Other: Visual Analog Scale (VAS); Behavioral: Impact of Event Scale - Revised (IES-R); Biological: Rectal swab sampling

INTERVENTIONS:
Other: Animal assisted therapy — Patients of AAT group will leave their hospital bedroom to go in the session room, where they will meet a dog, who has come with his veterinary student master. Animal assisted therapy session will last at most 20 minutes, in which the patient is going to interact with the dog, pet him, play with him, etc.
  Arms: Animal assisted therapy group
Biological: Nasal swab sampling — All patients will have nasal swab sampling at inclusion and 7 days after AAT session or sham session in order to screen multidrug resistant bacteria
Behavioral: STAI-Y and POMS Questionnaires — Before and after AAT or sham session, patients will answer State-Trait Anxiety Inventory Y (STAI-Y), Profile of Mood States (POMS) questionnaires.
Procedure: physiological parameters measure — Before and after AAT or sham session, blood pressure, heart rate dans respiratory rate will be measured.
Other: Visual Analog Scale (VAS) — Before and after AAT or sham session, pain will be evaluated thanks to VAS
Behavioral: Impact of Event Scale - Revised (IES-R) — Patients will answer IES-R questionnaire 3 months after AAT or sham session
Behavioral: satisfaction questionnaire — Patients of the AAT group will answer satisfaction questionnaire at the end of the AAT session and 3 months after AAT
  Arms: Animal assisted therapy group
Biological: Rectal swab sampling — All patients will have rectal swab sampling at inclusion and 7 days after AAT session or sham session in order to screen multidrug resistant bacteria

SUMMARY:
Assisted animal therapy (AAT) is getting more and more used worldwide, in such areas as gerontology, psychiatry, or oncology. It is a complementary therapy, and benefits for patients are various, including decrease of anxiety. In ICU, some case reports exist, but no study has ever been made in order to prove its benefits, not even its feasibility.

In ReAnimal, the investigator aims to compare a group of patients receiving assisted animal therapy, versus a group of patients not receiving it. Primary objective will be the evolution of anxiety scores between the 2 groups of patients. Secondary objectives will be the comparison of mood scores, post traumatic stress syndrome scores, pain scores, and physiologic parameters such as blood pressure, cardiac frequency. The investigating team will also compare multi drug resistant bacteria incidence between the 2 groups. In the assisted animal therapy group, patients will also be asked to answer a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in surgical ICU, not in acute stage of their ICU stay
* adult patient
* able to receive information and to give consent,
* with national social insurance

Exclusion Criteria:

* afraid of animal, dog phobia
* allergic to dog
* immunodepression (neutrophils <0.5 G/L), induced by treatment (chemotherapy, immunosuppressing treatment with high doses, corticotherapy for more than 2 weeks) or induced by disease (malignant blood disease, AIDS, transplantation, or splenectomy)
* sepsis ongoing
* patient known for having multidrug resistant bacteria
* wounds, or large bandages that could not correctly be covered, including external fixer
* central venous catheter, arterial catheter
* tracheostomy
* agitation, aggressiveness
* pregnant women
* patient deprived of freedom by juridical or administrative decision
* patient under legal protection measure
* patient receiving enforced psychiatric treatment
* patient admitted in a sanitary or social department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory Y (STAI-Y) score | Before randomization
  Self-administered questionnaire, of 20 questions whose answers are either "No", "Rather no" "Rather yes" "Yes". Points calculated are 1 point for each "No" answer, up to 4 points for each "Yes" answer. Thus, score can be at least 20 points, at most 80 points.
State-Trait Anxiety Inventory Y (STAI-Y) score | 2 days after inclusion, before AAT or sham session
  Self-administered questionnaire, of 20 questions whose answers are either "No", "Rather no" "Rather yes" "Yes". Points calculated are 1 point for each "No" answer, up to 4 points for each "Yes" answer. Thus, score can be at least 20 points, at most 80 points.
State-Trait Anxiety Inventory Y (STAI-Y) score | 2 days after inclusion, after AAT or sham session
  Self-administered questionnaire, of 20 questions whose answers are either "No", "Rather no" "Rather yes" "Yes". Points calculated are 1 point for each "No" answer, up to 4 points for each "Yes" answer. Thus, score can be at least 20 points, at most 80 points.

SECONDARY OUTCOMES:
Profile Of Mood States (POMS) score | 2 days after inclusion, before AAT or sham session
  Self-administered questionnaire, of 37 questions, whose answers are either "not at all", "a little", "moderately", "quite a lot", or "extremely". Each adjective in the POMS questionnaire is awarded the following score:
  * 0 - Not at all
  * 1 - A little
  * 2 - Moderately
  * 3 - Quite a Lot
  * 4 - Extremely except "Relaxed" and "Efficient" and they score the reverse:
  * 4 - Not at all
  * 3 - A little
  * 2 - Moderately
  * 1 - Quite a Lot
  * 0 - Extremely Thus, the score can range from 0 up to 148 points.
Profile Of Mood States (POMS) score | 2 days after inclusion, after AAT or sham session
  Self-administered questionnaire, of 37 questions, whose answers are either "not at all", "a little", "moderately", "quite a lot", or "extremely". Each adjective in the POMS questionnaire is awarded the following score:
  * 0 - Not at all
  * 1 - A little
  * 2 - Moderately
  * 3 - Quite a Lot
  * 4 - Extremely except "Relaxed" and "Efficient" and they score the reverse:
  * 4 - Not at all
  * 3 - A little
  * 2 - Moderately
  * 1 - Quite a Lot
  * 0 - Extremely Thus, the score can range from 0 up to 148 points.
Blood pressure | 2 days after inclusion, before AAT or sham session
  Physiological parameters noted on the patient usual monitoring in Intensive Care Unit (ICU), which the patient will keep during the whole session.
Blood pressure | 2 days after inclusion, after AAT or sham session
  Physiological parameters noted on the patient usual monitoring in Intensive Care Unit (ICU), which the patient will keep during the whole session.
Heart rate | 2 days after inclusion, before AAT or sham session
  Physiological parameters noted on the patient usual monitoring in Intensive Care Unit (ICU), which the patient will keep during the whole session.
Heart rate | 2 days after inclusion, after AAT or sham session
  Physiological parameters noted on the patient usual monitoring in Intensive Care Unit (ICU), which the patient will keep during the whole session.
Respiratory rate | 2 days after inclusion, before AAT or sham session
  Physiological parameters noted on the patient usual monitoring in Intensive Care Unit (ICU), which the patient will keep during the whole session.
Respiratory rate | 2 days after inclusion, after AAT or sham session
  Physiological parameters noted on the patient usual monitoring in Intensive Care Unit (ICU), which the patient will keep during the whole session.
Visual Analog Scale (VAS) score | 2 days after inclusion, before AAT or sham session
  Pain scale, from 0 = no pain at all, up to 10 = pain at maximum level
Visual Analog Scale (VAS) score | 2 days after inclusion, after AAT or sham session
  Pain scale, from 0 = no pain at all, up to 10 = pain at maximum level
Presence of Multi-drug resistant bacteria | At inclusion
  Nasal and rectal sampling, looking for methicillin resistant staphylococcus aureus in nasal sampling, and multi-drug resistant bacteria in rectal sampling
Presence of Multi-drug resistant bacteria | 7 days after AAT or sham session
  Nasal and rectal sampling, looking for methicillin resistant staphylococcus aureus in nasal sampling, and multi-drug resistant bacteria in rectal sampling
Impact of Event Scale - Revised (IES-R) score | 90 days after AAT or sham session
  Score for post traumatic stress disease. 22 questions self administered, whose answers are either "not at all", "a little", "moderately", "quite a lot", or "extremely". Each question is awarded score from 0 ("not at all") up to 4 ("extremely"). Thus, the total score ranges from 0 up to 88 points.
Patient Satisfaction score | 2 days after inclusion, at the end of AAT session
  Only for AAT group
Patient Satisfaction score | 90 days after AAT session
  Only for AAT group
Caregiver Satisfaction score | 2 days after inclusion, at the end of AAT session
Caregiver Satisfaction score | 90 days after AAT or sham session

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume PETIT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot - Anesthesiology department, Lyon, France